CLINICAL TRIAL: NCT02787239
Title: Clinical Study to Compare the Efficacy and Safety of Rituximab Biosimilar HLX01 and Rituximab in Combination With CHOP, in Previously Untreated Subjects With CD20+ DLBCL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HLX01-NHL03
Record Dates: First submitted 2016-05-18; First posted 2016-06-01 (Estimated); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: B-cell Non Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- HLX01 (Experimental): 375mg/m2 iv q3w, 6 cycles(each cycle is 3 weeks)
  Interventions: Drug: HLX01; Drug: CHOP
- Rituximab (Active Comparator): 375mg/m2 iv q3w, 6 cycles(each cycle is 3 weeks)
  Interventions: Drug: Rituximab; Drug: CHOP

INTERVENTIONS:
Drug: HLX01
  Arms: HLX01
Drug: Rituximab
  Arms: Rituximab
Drug: CHOP

SUMMARY:
Multicenter, Randomized, Double-blind, Parallel, Phase III Clinical Study to Compare the Efficacy and Safety of Rituximab Biosimilar HLX01 and MabThera in Combination With CHOP, in Previously Untreated Subjects With CD20+ DLBCL

ELIGIBILITY:
Inclusion Criteria:

* Untreated CD20-positive DLBCL confirmed.
* IPI score of 1 to 2, Stage I ~ IV, Score 0 needs to accompanied by bulky disease, which is defined as the presence of a tumor mass with a diameter of more than 7.5 cm.
* ECOG performance status of 0 to 2.
* More than 6 months life expectancy.
* At least one measurable lesion: For nodal tumor mass, more than 1.5 cm in the long axis and more than 1.0 cm in the short axis; For extranodal tumor mass, more than 1.0 cm in the long axis.
* 18 years to 70 years; Male or female patients.

Exclusion Criteria:

* Known allergic reactions against human or murine monoclonal antibody, murine products, or foreign proteins.
* Known allergic reactions against any component of CHOP regimen.
* Previous treatment for NHL, including chemotherapy, immunotherapy, partial radiotherapy for lymphoma, monoclonal antibody therapy or surgical treatment (excluding lymph node biopsies and surgical resection for non-lymphoma lesions).
* History of cytotoxic drugs treatment or anti-CD20 monoclonal antibody treatment for other disease (e.g., rheumatoid arthritis).
* Prior use of any monoclonal antibody within 3 months.
* Primary central nervous system(CNS) lymphoma, secondary CNS involvement, grey zone lymphoma (GZL) between burkitt and DLBCL, primary effusion lymphoma, plasmablastic lymphoma, primary cutaneous DLBCL, anaplastic lymphoma kinase(ALK) positive DLBCL or transformed lymphoma.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2015-10; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Overall Response Rate (ORR) | 18 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, China

REFERENCES:
- [Result] Shi Y, Song Y, Qin Y, Zhang Q, Han X, Hong X, Wang D, Li W, Zhang Y, Feng J, Yang J, Zhang H, Jin C, Yang Y, Hu J, Wang Z, Jin Z, Su H, Wang H, Yang H, Fu W, Zhang M, Zhang X, Chen Y, Ke X, Liu L, Yu D, Chen G, Wang X, Jin J, Sun T, Du X, Cheng Y, Yi P, Zhao X, Ma C, Cheng J, Chai K, Luk A, Liu E, Zhang X. A phase 3 study of rituximab biosimilar HLX01 in patients with diffuse large B-cell lymphoma. J Hematol Oncol. 2020 Apr 16;13(1):38. doi: 10.1186/s13045-020-00871-9. PMID 32299513
- See also: 286PFirst china-manufactured proposed rituximab biosimilar met primary efficacy and safety endpoints in CD20-positive diffuse large B-cell lymphoma (generics). Annals of Oncology 2018, 29 (suppl_9), mdy437.005-mdy437.005 — https://doi.org/10.1093/annonc/mdy437.005
- See also: A new population model validated pharmacokinetic similarity of HLX01 and rituximab in B-cell lymphoma. Annals of Oncology 2019, 30. — https://doi.org/10.1093/annonc/mdz251.015
- See also: 266OA population pharmacokinetic model: Assessment of pharmacokinetic similarity of HLX01 and rituximab in diffuse large B-cell lymphoma. Annals of Oncology 2019, 30 (suppl_9), mdz427. — https://doi.org/10.1093/annonc/mdz427